CLINICAL TRIAL: NCT02805283
Title: Direct to Patient Survey to Examine Treatment Satisfaction and Experience With Dapagliflozin Compared to Sulfonylureas
Brief Title: Dapagliflozin Patient Satisfaction Survey
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Optum, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: D1690R00026
Record Dates: First submitted 2016-06-02; First posted 2016-06-20 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dapagliflozin, dapagliflozin/met ER: Dapagliflozin cohort have at least one pharmacy claim for either dapagliflozin or dapagliflozin/metformin ER in the most recent month of pharmacy data and no pharmacy claims for a medication in the same drug class during the 6 months prior to sample identification.
- Sulfonylurea: Sulfonylurea cohort have at least one pharmacy claim for sulfonylurea in the most recent month of pharmacy data and no pharmacy claims for a medication in the same drug class during the 6 months prior to sample identification.

SUMMARY:
The purpose of this study is to evaluate the diabetes related treatment satisfaction for patients with type 2 diabetes mellitus

DETAILED DESCRIPTION:
This is a cross-sectional, observational patient survey study. Study subjects will be adult commercial members of the large US health plan affiliated with Optum with evidence of T2D initiating dapagliflozin or a sulfonylurea medication within the 3 months prior to survey mailing.

ELIGIBILITY:
Inclusion Criteria:

* At least one pharmacy claim for dapagliflozin or dapagliflozin/metformin ER in the most recent month of pharmacy data and no pharmacy claims for an SGLT2 medication during the 6 months prior to sample identification.
* Evidence of T2D diagnosis.
* Age ≥18 as of the drug index date.
* 6 months of continuous enrollment in a commercial health plan with both pharmacy and medical benefits during the identification period through the patient interview sample identification date.
* Self-reported T2D diagnosis during the patient interview.

Exclusion Criteria:

* Patients with evidence of type 1 diabetes mellitus and unknown type
* Patients who are pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 Diabetes patients with administrative claims data from Optum Research Database (US Commercial Claims Data)
Sampling Method: Non-Probability Sample
Enrollment: 653 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Condition-specific treatment satisfaction | 2 weeks
  Condition-specific treatment satisfaction as measured by the Diabetes Treatment Satisfaction Questionnaire (DTSQ)

SECONDARY OUTCOMES:
Medical Outcomes Study (MOS) Short Form Health Survey SF-12 or SF-36 | 4 weeks
  MOS Short Form Health Survey SF-12 or SF-36
Morisky Medication Adherence Scale | 1 month
  Medication adherence
Hypoglycemia Fear Survey | 4 weeks
  Fear of hypoglycemia (HFS)
Self-reported body weight | 1 month
  Self-reported body weight

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Bell, PharmD, MSPhr, Study Chair — AstraZeneca
Locations (1):
- Reasearch Site, Eden Prairie, Minnesota, United States